CLINICAL TRIAL: NCT04777838
Title: Effectiveness of the Use of Antidepressants in the Treatment of Muscle Type Temporomandibular Disorders
Brief Title: Myofascial Pain Patients' Response to the Administration of Low Doses of Amitriptyline and Citalopram Compared With the Use of Bite Splint
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Coimbra (Other)
Collaborators: Instituto de Investigación Biomédica de Salamanca (Other)
Responsible Party: Principal Investigator, Bruno Macedo de Sousa, Principal Investigator, University of Coimbra
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADP2021
Record Dates: First submitted 2021-02-10; First posted 2021-03-02 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-03

CONDITIONS: Muscle Type Temporomandibular Disorders; Myofascial Pain of the Masticatory Muscles
MeSH Terms: interventions — Citalopram; Amitriptyline; Occlusal Splints

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Citalopram (Active Comparator): Citalopram 10mg
  Interventions: Drug: Citalopram 10 MG
- Amitriptyline (Active Comparator): Amitritptyline 25 mg
  Interventions: Drug: Amitriptyline
- Bite Splint (Active Comparator): Michigan Splint, nocturnal use
  Interventions: Device: Bite Splint

INTERVENTIONS:
Drug: Citalopram 10 MG — 10 mg of citalopram every day
  Arms: Citalopram
Drug: Amitriptyline — 25mg of Amitriptyline every
  Arms: Amitriptyline
Device: Bite Splint — Night use of occlusal splint
  Arms: Bite Splint

SUMMARY:
The aim of this study is evaluate the effectiveness of the use of antidepressants in the treatment of muscle type temporomandibular disorders, with a sample of 60 to 80 participants.

DETAILED DESCRIPTION:
Temporomandibular Disorders (TMDs) involve alterations of the temporomandibular joint (TMJ), masticatory muscles, and related structures.

Epidemiologic data indicates that 33% of the general population has at least one symptom of a temporomandibular disorder (TMD) and 6% to 7% have TMDs severe enough to seek specific treatment.

The etiology of pain and disability in myofascial pain is understood via a bio- psychosocial model reflecting a complex interaction between physical, behavioral, social, and psychological factors. In turn, the treatment of myofascial pain is often multimodal.

Ongoing pain may be associated with co-morbid conditions such as anxiety, depression and sleeplessness. It is important to recognize and treat emotional distress as well as physical symptoms. Chronic pain and depression seem to share common neurochemical substrata and perhaps even similar dysfunctional alterations.

Chronic syndromes such as bruxism and TMD are commonly associated with depression. Research Investigator reported that 39% of patients with TMD are moderately to severely depressed and 55% have moderate to severe somatization symptoms. A cross-cultural study by List and Dworkin supported these findings, showing that 45% of Swedish patients and 51% of American patients who met the diagnostic criteria for TMD also suffered from moderate to severe depression.

If pain assumes a chronic nature, more centrally mediated mechanisms take effect, for which peripherally acting analgesics have less efficacy. The clinician must recognize the involved alterations in pain characteristics, such as quality, duration, and intensity, as peripheral pain becomes more continuous, diffuse, and difficult to localize. In such instances, the possibility of new targets for treatment emerges.

The prominence of tryciclic antidepressants (TCAs) as a first-line treatment has declined over time and the introduction of more tolerable medications such as the selective serotonin reuptake inhibitors (SSRIs) has been done. TCAs are still used today, but they are most commonly prescribed for patients whose depression does not respond to SSRIs or serotonin and norepinephrine reuptake inhibitors (SNRIs). TCAs are also used to treat depressed patients with somatization pain or insomnia, due to their low addictive risk and sedative and analgesic qualities; however, TCAs are associated with a high suicide risk when taken in overdose.

For the past several years, tricyclic antidepressants have been used successfully to manage and control a variety of chronic pain conditions. Research Investigators reported that a pharmacological protocol for the control of pain associated with chronic temporomandibular disorders (TMD) based on the use of amitriptyline and found that 25 mg/day of amitriptyline was sufficient to significantly reduce the pain of chronic TMD without producing side effects.

Research Investigator showed that 75 mg of amitriptyline provided significantly more pain relief than 25 or 50mg in patients with chronic pain. However, the patients on higher doses also had more adverse events such as dry mouth and drowsiness. It should also be kept in mind that no dose-response relation- ship has been demonstrated for the antidepressant or mood effects of amitriptyline.

Research Investigator compared the effectiveness of cognitive behavioral therapy (CBT) and amitriptyline in combination and separately in patients with chronic TMD. They discovered improvements in all subgroups (CBT alone, amitriptyline alone, CBT plus amitriptyline, and the placebo group) with an average decrease in pain intensity of 55%. The combination group of CBT plus amitriptyline, however, was the only group that continued to show improved scores on the visual analog pain scale at the follow-up 4 weeks after treatment was completed.

The neurotransmitter serotonin regulates a wide range of functions including sleep, temperature, and mood. Based on that we could suggest that it has a positive impact on Chronic Pain patients. However, Serotonin also suppresses dopamine release from the mesocortical tract, which can result in serotonin-induced disinhibition of movement. In other words, dopamine functions to prevent spontaneous movements, but if serotonin inhibits the action of dopamine, then spontaneous movements can occur. This is thought to be one of the most plausible mechanisms involved in the repetitive muscle contractions seen in bruxism. This mechanism also explains how the SSRIs, which increase concentrations of serotonin, have the ability to deregulate movement and induce bruxism.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated at the Centro Hospitalar e Universitário de Coimbra (CHUC);
* Patients who, according to the diagnostic Criteria for Temporomandibular disorder (DC/TMD) , present Myofascial pain in the masticatory muscles for more than 6 months;
* Adult patients

Exclusion Criteria:

* Under 18 years old;
* Pregnants,
* Patients who have related adverse effects to the citalopram and/or amitriptyline;
* Patients presenting severe diseases like coronary pathology, renal insufficiency, active cancer, respiratory insufficiency;
* Patients who have been treated to myofascial pain before

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 3 weeks
  Pain intensity according to a visual analogue scale from 0 to 10.
Pain intensity | 6 weeks
  Pain intensity according to a visual analogue scale from 0 to 10.
Pain intensity | 9 weeks
  Pain intensity according to a visual analogue scale from 0 to 10.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno M Sousa, Principal Investigator — Institute for Occlusion and Orofacial Pain Faculty of Medicine, University of Coimbra
Locations (1):
- CHUC - Centro Hospitalar e Universitário de Coimbra, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: Undecided